CLINICAL TRIAL: NCT02334033
Title: Cystatin C and Uncontrolled Hypertension
Status: Completed | Type: Observational
Sponsor: Ankara University (Other)
Responsible Party: Principal Investigator, Özgür Ulaş Özcan, MD, Ankara University
Other Study IDs: AnkaraUHyper
Record Dates: First submitted 2015-01-02; First posted 2015-01-08 (Estimated); Last update posted 2015-01-27 (Estimated); Status verified 2015-01

CONDITIONS: Uncontrolled Hypertension
Keywords: hypertension; blood pressure; cystatin C; real-life; kidney
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional

INTERVENTIONS:
Other: other

SUMMARY:
Hypertension is an underdiagnosed and undertreated disease in real-life. Blood pressure and kidney functions are known to be closely related. Increased serum level of Cystatin C, a sensitive biomarker for renal function, seems to predict adverse cardiovascular events. The investigators aimed to evaluate the predictive value of serum Cystatin C for control of hypertension in a community-based study.

ELIGIBILITY:
Inclusion Criteria:

* Individuals who accept to participate to the survey
* > 18 years

Exclusion Criteria:

* Individuals who are not able to complete the questionnaire
* Individuals who didn't give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults residing in both rural and urban communities
Sampling Method: Non-Probability Sample
Enrollment: 903 (Actual)
Dates: Start 2014-01; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
The prevalence of uncontrolled hypertension | At subject enrollment
  The outcome measures will be obtained at the time of enrollment

SECONDARY OUTCOMES:
The value of cystatin C to determine uncontrolled hypertension | At subject enrollment
  The outcome measures will be obtained at the time of enrollment

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara University School Of Medicine, Department of Cardiology, Ankara, Turkey (Türkiye)